CLINICAL TRIAL: NCT00942981
Title: Functional Relevance of Dopamine Receptors in Healthy Controls and Patients With Schizophrenia: Characterization Through [11C]NNC-112 and [18F]Fallypride Positron Emission Tomography
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090176; 09-M-0176
Record Dates: First submitted 2009-07-18; First posted 2009-07-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-20

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: PET Study; (18F) Fallypride; (11C)NNC-112; D-1 Receptors; Schizophrenia; Natural History; Schizoaffective Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: healthy volunteers
  Interventions: Drug: PET
- patients: patients with schizophrenia, schizoaffective disorder or other psychotic disorders aged18-60
  Interventions: Drug: PET

INTERVENTIONS:
Drug: PET — Brain dopamine D1 and D2/3 receptor regional binding potentials measured by [11C]NNC-112 and [18F]Fallypride PET.

SUMMARY:
Background:

* Some illnesses, such as schizophrenia, have effects on brain cells called dopamine receptors, which are required for normal brain function. People with schizophrenia have difficulty thinking and experience hallucinations and delusions. Medications that change brain dopamine receptors can decrease these hallucinations and delusions.
* The cause of schizophrenia and its association with brain dopamine receptors is not known but may be clarified by studying dopamine receptors in people who have dopamine disorders (such as schizophrenia) and those who do not. Researchers are interested in studying the dopamine system to gain a better idea of how dopamine disorders develop, which may lead to better medical care for people with schizophrenia.

Objectives:

- To study the amount and distribution of two types of dopamine receptors.

Eligibility:

* Individuals between the ages of 18 and 60 who have schizophrenia.
* Healthy volunteers between the ages of 18 and 90.

Design:

* Participants will undergo a full screening, with physical and psychological history, a neurological examination, and blood and urine samples.
* Participants will have a blood flow map of the brain recorded with a positron emission tomography (PET) brain scan. A magnetic resonance imaging (MRI) scan will also be performed to determine brain anatomy.
* To study the amount and distribution of dopamine receptors in the brain, participants will receive a small amount of a radioactive chemical in the vein, followed by a PET scan.
* The procedure will be performed twice in two separate sessions, once for [18F]fallypride and once for [11C]NNC-112.

DETAILED DESCRIPTION:
OBJECTIVES

Dopaminergic (DA) modulation of brain function is disturbed in several disabling psychiatric disorders and represents the target of key psychopharmacologic agents, such as neuroleptics. Schizophrenia has been considered a prototype of dysregulated DA signaling, with associated prefrontal cortex (PFC) dysfunction. Prevailing views attribute key symptoms of schizophrenia to deficient DA signaling within mesocortical DA tracts. Little is known, however, about the pre-, intra-, and post-synaptic processes that contribute to dopaminergic dysregulation. Regional cortical DA activity, critical to these processes, has been difficult to measure in patients with the available imaging techniques. The current clinical study aims to address this open issue by taking advantage of two recently developed positron emission tomography (PET) radioligands, [(11)C]NNC-112 and [(18)F]Fallypride, that bind differentially and with a higher binding potential (BP) than previous compounds to the D(1) (NNC-112) or D(2/3) (fallypride) receptors. By measuring the regional BP of these two compounds, cortical and subcortical DA receptor anomalies will be characterized in schizophrenia. Within the Clinical and Translational Neuroscience Branch (CTNB), this PET protocol is expected to add crucial information about DA receptor status to ongoing regional cerebral blood flow (rCBF), magnetic resonance imaging (MRI), magneto-encephalography (MEG) and genetic studies. It will lead to an improved understanding of the modulatory influence of DA on frontal lobe functioning and facilitate the study of how genetic polymorphisms interact with regional changes in D(1) and D(2/3) receptors to increase the risk for schizophrenia.

Some specific hypotheses to be tested are as follows:

D1 BP in frontal cortex will be affected by age, elevated in schizophrenia and inversely correlated with cognitive performance in patients and healthy controls.

Cortical D2/3 receptor BP will be affected by age and inversely correlated with performance on tests of frontal lobe function in patients and healthy controls.

Striatal D2/3 receptor BP will be altered in patients.

Polymorphisms in the catechol-O-methyl transferase (COMT), D1 and D2 genes as well as other schizophrenia risk genes will affect DA receptor BP in frontal cortex.

The ratio of cortical D1 and D2/3 receptor BPs will be affected by age and related to risk for schizophrenia, cognitive performance and polymorphisms in the COMT gene and other schizophrenia risk genes

STUDY POPULATION

It will include 100 patients with schizophrenia, schizoaffective disorder or other psychotic disorders aged 18-60, and 230 healthy controls, aged 18-90. Fifty of the controls will be matched to the patients by age and sex.

DESIGN

Dopamine D(1) and D(2/3) receptor regional binding potentials (BP) will be quantified by PET in medication-free patients and controls. High resolution T1-weighted magnetic resonance imaging (MRI) scans will be obtained for co-registration purposes. Additionally, through enrollment in other ongoing protocols (00-M-0085, 90-M-0014, 01-M-0232, 95-M-0150, 89-M-0160), rCBF, functional MRI, cognitive and genetic data will be obtained and compared with D(1) and D(2/3) receptor BP data obtained from this protocol.

OUTCOME MEASURES

Brain dopamine D(1) and D(2/3) receptor regional binding potentials measured by [[(11)C]NNC-112 and [(18)F]Fallypride PET.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects will be recruited among individuals volunteering for NIH protocol 95-M-0150 A Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings (PI: Karen Berman, M.D.), NIH protocol 00-M-0085 Structural and Functional Imaging of Neuropsychiatric Patients and Normal Volunteers with 3.0 Tesla MRI and Magnetoencephalography. (P.I.: Karen Berman, MD) or NIH protocol 89-M-0160 "Inpatient Evaluation of Neuropsychiatric Patients" (PI: Daniel Eisenberg, M.D.). Most included patients, with schizophrenia, schizoaffective disorder or other non-excluded psychotic disorders, will be managed on the NIMH inpatient ward for the duration of their participation.
* Only adult subjects who are able to provide informed consent will be studied.
* Patients will be between 18 and 60 years of age. Healthy controls will be matched by age and sex to the patients. In addition, to study age effect on DA receptors, healthy controls will be included up to the age of 90 years.
* Control subjects must be healthy based on history, laboratory and physical exam obtained through the above mentioned protocols.

EXCLUSION CRITERIA:

-Subjects will be excluded if they don t fit the study requirements regarding age, ability to provide informed consent, absence of significant general medical, neurological or psychiatric disorders (except the disorder object of study), or intake of substances that

interfere with central dopaminergic signaling.

* NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.
* Pregnant or breast feeding
* Current psychiatric illness except for patients with schizophrenia, schizoaffective disorder or other psychotic disorder
* Secondary causes of schizophrenia-like syndromes, e.g. amphetamine abuse, brain infarction, tumor, or trauma
* Neurological disorders except those of exclusively peripheral location
* Current or prior use (within 4 weeks) of substances that interfere with central dopaminergic signaling (e.g. antipsychotics, dopamine receptor agonists, anticholinergics, MAO-B inhibitors)
* History of any (excepting nicotine- related) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).
* Cumulative lifetime history of any (excepting nicotine -related) DSM5-defined mild substance use disorder (or any DSM-IV-defined substance abuse), either in excess of 5 years total or not in remission for at least 6 months.
* Severe systemic disease, such as hypothyroidism not compensated by medication
* Laboratory tests with clinically significant abnormalities
* History of a significantly abnormal EEG, cranial CT or MRI
* Conditions that increase risk for MRI (pacemaker devices, ferromagnetic metal implants, etc.)
* Prior participation in other research protocols such that radiation exposure would exceed the annual NIH RSC limits
* Any medical condition that in the opinion of the investigators would interfere with the safe conduct of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It will include 100 patients with schizophrenia, schizoaffective disorder or other psychotic disorders aged 18-60, and 230 healthy controls, aged 18-90.
Sampling Method: Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2009-11-13 (Actual)

PRIMARY OUTCOMES:
Brain dopamine D1 and D2/3 receptor regional binding potentials | ongoing
  Brain dopamine D1 and D2/3 receptor regional binding potentials

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Berman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ianni AM, Eisenberg DP, Boorman ED, Constantino SM, Hegarty CE, Gregory MD, Masdeu JC, Kohn PD, Behrens TE, Berman KF. PET-measured human dopamine synthesis capacity and receptor availability predict trading rewards and time-costs during foraging. Nat Commun. 2023 Sep 30;14(1):6122. doi: 10.1038/s41467-023-41897-0. PMID 37777515
- [Derived] Hegarty CE, Ianni AM, Kohn PD, Kolachana B, Gregory M, Masdeu JC, Eisenberg DP, Berman KF. Polymorphism in the ZNF804A Gene and Variation in D1 and D2/D3 Dopamine Receptor Availability in the Healthy Human Brain: A Dual Positron Emission Tomography Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Jan;8(1):121-128. doi: 10.1016/j.bpsc.2020.12.006. Epub 2021 Mar 9. PMID 33712377
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-M-0176.html